CLINICAL TRIAL: NCT02818387
Title: The Effect of Remifentanil and Midazolam on Propofol for Loss of Consciousness During Induction of Anesthesia in Elderly Patients
Brief Title: Remifentanil and Midazolam on Propofol for Loss of Consciousness in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jiwon An, MD, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3-2015-0222
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia
Keywords: propofol; midazolam; remifentanil; combination; synergic; pharmacodynamics; Loss of consciousness
MeSH Terms: conditions — Unconsciousness | interventions — Propofol; Remifentanil; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group P (Active Comparator): Induction with propofol bolus. Dose will be started at 0.5 mg/kg and will be adjusted as described in summary.
  Interventions: Drug: Propofol
- Group PR (Active Comparator): Induction with propofol and remifentanil. Remifentanil infusion 0.125 mcg/kg/min for 5 min followed by propofol bolus Propofol dose will be started at 0.5 mg/kg and will be adjusted as described in summary.
  Interventions: Drug: Propofol; Drug: Remifentanil
- Group PMR (Active Comparator): Induction with propofol, midazolam and remifentanil. Remifentanil infusion 0.125 mcg/kg/min for 5 min followed by midazolam 0.015 mg/kg bolus 1 min after remifentanil infusion start and propofol bolus administration.
  Propofol dose will be started at 0.5 mg/kg and will be adjusted as described in summary.
  Interventions: Drug: Propofol; Drug: Remifentanil; Drug: Midazolam

INTERVENTIONS:
Drug: Propofol — Propofol bolus dose administration according to the predetermined dose by biased coined design up-and-down study.
  Other Names: Fresofol
Drug: Remifentanil — Remifentanil 0.125 mcg/kg/min infusion for 5 min before propofol administration.
  Other Names: Ultiva
  Arms: Group PMR; Group PR
Drug: Midazolam — Remifentanil 0.125 mcg/kg/min infusion for 5 min before propofol administration followed by midazolam 0.015 mg/kg administration 1 min after remifentanil infusion start.
  Arms: Group PMR

SUMMARY:
Propofol is a well-known induction agent which can provide sound and quick hypnosis with anti-emetic effects. However, dose dependent hypotension or bradycardia have reported while using this agent. Propofol in combination with remifentanil or midazolam can result in synergistic or additive effect in elderly patients. There are not many studies which provide minimum dose of propofol to induce hypnosis in combination with these agents and advantage of the combination.

The elderly patients (over 65 years old) who are scheduled to undergo general anesthesia are enrolled in this study. 120 patients will be randomly allocated to 3 groups(P, PR, PMR). Sample size have been decided due to the previous studies which have mentioned 40 participants as a adequate sample size for this biased coin design - up and down study.

After receiving informed consent, patients will be participated in this study. No premedication will be given to the patients before induction. The patients in group P will receive general anesthesia only with propofol and group PR and PMR will receive 0.125 mcg/kg/min remifentanil infusion for 5 min prior to propofol administration. The patients in group PMR will receive 0.015 mg/kg bolus dose of midazolam 1 min after the start of the remifentanil infusion. Initial propofol dose will be 0.5 mg/kg in each group and the dose will be changed by the result of prior study participant.

'Success' of this study will be defined as loss of both verbal response and eyelash reflex in 3 min after propofol administration. When 'success', the next patient will receive the same dose(in 18/19 probability) or 0.125 mg/kg lower dose(in 1/19 probability) of propofol. When 'failure', the next patient will receive 0.125 mg/kg higher dose of propofol at induction period.

DETAILED DESCRIPTION:
Propofol is a well-known induction agent which can provide sound and quick hypnosis with anti-emetic effects. However, dose dependent hypotension or bradycardia have reported while using this agent. Propofol in combination with remifentanil or midazolam can result in synergistic or additive effect in elderly patients. There are not many studies which provide minimum dose of propofol to induce hypnosis in combination with these agents and advantage of the combination.

The elderly patients (over 65 years old) who are scheduled to undergo general anesthesia are enrolled in this study. 120 patients will be randomly allocated to 3 groups(P, PR, PMR). Sample size have been decided due to the previous studies which have mentioned 40 participants as a adequate sample size for this biased coin design - up and down study.

After receiving informed consent, patients will be participated in this study. No premedication will be given to the patients before induction. The patients in group P will receive general anesthesia only with propofol and group PR and PMR will receive 0.125 mcg/kg/min remifentanil infusion for 5 min prior to propofol administration. The patients in group PMR will receive 0.015 mg/kg bolus dose of midazolam 1 min after the start of the remifentanil infusion. Initial propofol dose will be 0.5 mg/kg in each group and the dose will be changed by the result of prior study participant.

'Success' of this study will be defined as loss of both verbal response and eyelash reflex in 3 min after propofol administration. When 'success', the next patient will receive the same dose(in 18/19 probability) or 0.125 mg/kg lower dose(in 1/19 probability) of propofol. When 'failure', the next patient will receive 0.125 mg/kg higher dose of propofol at induction period.

ELIGIBILITY:
Inclusion Criteria:

* The elderly patients (over 65 years old) who are scheduled to undergo general anesthesia.

Exclusion Criteria:

* ASA class (American Society of Anesthesiologist physical status classification) IV or higher
* Patients with history of allergy or side effects on propofol, remifentanil, midazolam
* BMI (body mass index) less than 20 or higher than 30
* Patients taking sedatives or hypnotic agents.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Loss of verbal response and eyelash reflex | 3 minutes after propofol administration
  Checking verbal response by verbal stimulation (response or no response).
Loss of eyelash reflex | 3 minutes after propofol administration
  Checking reflex by palpation of the levator palpebrae (reflex or no reflex).

SECONDARY OUTCOMES:
Mean blood pressure | baseline, propofol administration time (Just after finishing monitoring on the patient in P group, 5 minutes after remifentanil infusion start in PR and PMR group), 1 minute, 2 minutes and 3 minutes after propofol administration
  To compare differences among groups in mean blood pressure change (mmHg)
Heart rate | baseline, propofol administration time (Just after finishing monitoring on the patient in P group, 5 minutes after remifentanil infusion start in PR and PMR group), 1 minute, 2 minutes and 3 minutes after propofol administration
  To compare differences among groups in heart rate change (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, MD,PhD, Study Chair — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, Korea, South Korea

REFERENCES:
- [Background] Conway DH, Hasan SK, Simpson ME. Target-controlled propofol requirements at induction of anaesthesia: effect of remifentanil and midazolam. Eur J Anaesthesiol. 2002 Aug;19(8):580-4. doi: 10.1017/s0265021502000935. PMID 12200947